CLINICAL TRIAL: NCT01386333
Title: A Phase I Dose Finding Study of Intranasal Oxytocin in Frontotemporal Dementia, Protocol # FTDOXY10EF
Brief Title: Safety Study of Intranasal Oxytocin in Frontotemporal Dementia
Acronym: FTDOXY10EF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Consortium of Canadian Centres for Clinical Cognitive Research (Other)
Responsible Party: Principal Investigator, Elizabeth Finger, Cognitive Neurologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-11-232; 17783 (Other: REB)
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Frontotemporal Dementia
Keywords: Frontotemporal Dementia; oxytocin; Pick's disease
MeSH Terms: conditions — Frontotemporal Dementia; Pick Disease of the Brain | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oxytocin 24IU (Experimental): Oxytocin 24 IU administered intranasally twice daily for 1 week
  Interventions: Drug: oxytocin
- Oxytocin 48 IU (Experimental): 48 IU of intranasal oxytocin administered twice daily for 1 week
  Interventions: Drug: oxytocin
- 72 IU oxytocin (Experimental): 72 IU of intranasal oxytocin administered twice daily for 1 week
  Interventions: Drug: oxytocin
- Saline nasal spray (Placebo Comparator)
  Interventions: Drug: oxytocin; Drug: Saline Nasal Mist

INTERVENTIONS:
Drug: oxytocin — Patients will be randomized to receive intranasal oxytocin or placebo in a dose escalation paradigm with three dose cohorts: 24IU, 48IU and 72IU of intranasal oxytocin twice daily for 1 week
Drug: Saline Nasal Mist — Placebo arm wil receive saline nasal mist sprays matched in number to oxytocin dose cohorts
  Arms: Saline nasal spray

SUMMARY:
Oxytocin is a hormone produced by the brain that appears to have important roles in social cognition and emotion in humans. In a pilot study, the effects of a single dose of oxytocin on measures of emotion recognition and behaviour in patients with Frontotemporal Dementia were investigated. The results from the pilot study suggested that oxytocin may be associated with a modest improvement in neuropsychiatric behaviours seen in patients with Frontotemporal Dementia. To further examine the safety and tolerability of oxytocin in this disorder, the present study will examine the safety and tolerability of three different doses of intranasal oxytocin administered to patients with Frontotemporal Dementia twice daily for 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years
* Meets "Neary criteria" for diagnosis of probable frontotemporal dementia
* Neuroimaging (CT, MRI or SPECT scan) supports diagnosis of frontotemporal dementia
* Provides written informed consent and has a caregiver or legally acceptable representative who provides written informed consent.

Exclusion Criteria:

* Has a history of a myocardial infarction within the last two years or congestive heart failure.
* Current uncontrolled hypertension
* Current bradycardia (rate < 50 beats per minute/bpm) or tachycardia (rate > 100 bpm)
* Current hyponatremia
* Current use of prostaglandin medications
* Females who are pregnant or breastfeeding
* Use of any investigational or experimental drug or device within the last 60 days prior to screening or within 5 half-lives of the experimental drug , whichever is longer.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 week
  Safety and Tolerability of 24 international units (IU), 48 IU and 72 IU of intranasal oxytocin administered twice daily for 1 week to patients with Frontotemporal Dementia as assessed by the number of participants with adverse events. Adverse events will be assessed by a standardized questionnaire and serum sodium levels will be monitored.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory | 1 week
  Behavioural ratings at baseline and 1 week of oxytocin treatment compared to 1 week of placebo treatment
Frontal Behavioural Inventory | 1 week
Clinicians Global Impression of Change | 1 week
Clinical Dementia Rating- Frontotemporal Lobar Degeneration | 1 week
Interpersonal Reactivity Index | 1 week
Multi-faceted Empathy Test | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Finger, MD, Principal Investigator — University of Western Ontario, Lawson Health Research Institute
Locations (1):
- Cognitive Neurology and Alzheimer Research Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Finger EC, MacKinley J, Blair M, Oliver LD, Jesso S, Tartaglia MC, Borrie M, Wells J, Dziobek I, Pasternak S, Mitchell DG, Rankin K, Kertesz A, Boxer A. Oxytocin for frontotemporal dementia: a randomized dose-finding study of safety and tolerability. Neurology. 2015 Jan 13;84(2):174-81. doi: 10.1212/WNL.0000000000001133. Epub 2014 Dec 10. PMID 25503617